CLINICAL TRIAL: NCT00003734
Title: A Randomised Comparison of Short and Protracted Neoadjuvant Hormonal Therapy Prior to Radiation Therapy of High Risk Localized Prostate Cancer
Brief Title: Combination Hormone Therapy Followed by Radiation Therapy in Treating Patients With Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Luke's Hospital, Ireland (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066849; ICORG-97-01; EU-98060
Record Dates: First submitted 1999-11-01; First posted 2003-12-09 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2011-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Triptorelin Pamoate; Radiotherapy

INTERVENTIONS:
Drug: flutamide
Drug: triptorelin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using triptorelin and flutamide may fight cancer by reducing the production of androgens. It is not yet known whether giving hormone therapy for 4 months is more effective than giving therapy for 8 months prior to radiation therapy for prostate cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of combination hormone therapy for 4 or 8 months followed by radiation therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of 4 months vs 8 months of luteinizing hormone-releasing hormone (LHRH) agonist therapy combined with antiandrogen therapy prior to radiotherapy, in terms of disease-free survival and overall survival, in patients with stage I-IV localized invasive prostate cancer.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms. All patients receive triptorelin IM once a month and oral flutamide three times daily with meals. Patients randomized to arm I receive this therapy regimen for 4 months. Patients randomized to arm II receive this therapy regimen for 8 months. All patients then undergo radiotherapy 5 days a week for 7 weeks within 2 months of the last injection of triptorelin and within 1 month of the last oral flutamide tablet. Patients are followed every 3 months after radiotherapy.

PROJECTED ACCRUAL: A total of 276 patients (138 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed invasive adenocarcinoma of the prostate Stage I or II (PSA greater than 20 or Gleason score at least 7) OR Stage III or IV (any PSA, any Gleason) Histologically confirmed benign nodal status No distant metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other prior malignancy except nonmelanoma skin cancer No other uncontrolled illness that would prevent compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No prior or other concurrent hormonal therapy Radiotherapy: Not specified Surgery: No prior treatment other than transurethral prostatectomy No prior orchiectomy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: John Gerard Armstrong, MD, MB, MRCPI, Study Chair — Saint Luke's Hospital
Locations (12):
- Ireland (11):
  - Cork University Hospital, Cork
  - Letterkenny Hospital, Donnegal
  - St. Vincent's Hospital, Dublin
  - Saint Luke's Hospital, Dublin
  - Mater Misericordiae Hospital, Dublin
  - Adelaide and Meath Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Bon Secours Hospital, Galway
  - Galway University Hospital, Galway
  - Regional Hospital - Limerick, Limerick
  - Sligo General, Sligo
- Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Result] Armstrong JG, Gillham CM, Dunne MT, Fitzpatrick DA, Finn MA, Cannon ME, Taylor JC, O'Shea CM, Buckney SJ, Thirion PG. A randomized trial (Irish clinical oncology research group 97-01) comparing short versus protracted neoadjuvant hormonal therapy before radiotherapy for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2011 Sep 1;81(1):35-45. doi: 10.1016/j.ijrobp.2010.04.065. Epub 2010 Aug 25. PMID 20797824